CLINICAL TRIAL: NCT02901782
Title: Personalized Titanium Plate Improves Clinical Outcome in Microwave Ablation of Bone Tumors Around the Knee
Brief Title: The Application of Personalized Titanium Plate in the Bone Tumors Around the Knee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou General Hospital of Guangzhou Military Command (Other)
Collaborators: Medical Center of Assessment, Prevention and Treatment of Bone & Joint Diseases, Guangdong, China (Other); The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Yu Zhang, Principal Investigator, Clinical Professor, Guangzhou General Hospital of Guangzhou Military Command
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GuangzhouGH002
Record Dates: First submitted 2016-08-31; First posted 2016-09-15 (Estimated); Last update posted 2017-02-13 (Actual); Status verified 2017-02

CONDITIONS: Bone Tumors
Keywords: Knee; Titanium Plate
MeSH Terms: conditions — Bone Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Personalized titanium plate (Experimental): Ten males and two females with a mean age of 22.8 years were recruited. They all had bone tumor around the knee.
  Interventions: Procedure: Personalized titanium plate

INTERVENTIONS:
Procedure: Personalized titanium plate — 3D models of tumor-bearing bone segments were constructed by using computed tomography (CT) and magnetic resonance imaging (MRI). The 3D models were used to design the model of personalized titanium plates. The model of the plates was transferred into a numerical control machine for manufacturing the personalized titanium plates by 3D printing technology. The plates were then surgically implanted for reconstruction assistance following microwave-induced hyperthermia to remove the bone tumor. Implementation parameters and knee function were then evaluated.

SUMMARY:
Microwave ablation of bone tumors is time-consuming and usually results in postoperative fractures. Hence the investigators designed and fabricated a titanium plate customized to the patient's bone structures for fixation after the removal of tumorous tissue, to improve the clinical outcomes of microwave ablation.

DETAILED DESCRIPTION:
3D models of tumor-bearing bone segments were constructed by using computed tomography (CT) and magnetic resonance imaging (MRI). The 3D models were used to design the model of personalized titanium plates. The model of the plates was transferred into a numerical control machine for manufacturing the personalized titanium plates by 3D printing technology. The plates were then surgically implanted for reconstruction assistance following microwave-induced hyperthermia to remove the bone tumor. Implementation parameters and knee function were then evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of primary malignant bone tumors in the distal femur or proximal tibia according to the preoperative biopsy.
2. Malignant soft tissue tumor invading distal femur or proximal tibia.
3. The patients have the opportunity of limb salvage and treatment of microwave-induced hyperthermia in situ and reconstruction with internal fixation.

Exclusion Criteria:

1. Distant metastasis.
2. Benign tumor.
3. Metastatic tumor around the knee.
4. No indication of limb salvage.
5. Malignant soft tissue tumor without bone invasion.
6. Recrudescent tumors.

Ages: 5 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-01; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Musculoskeletal Tumor Society score | An average of 29 months
Mean maximum flexion of the knee | An average of 29 months
The six degrees of freedom of the gait | An average of 29 months
  including flexion/extension, adduction/abduction, internal/external rotation, anteroposterior translation, distal/lateral translation, medial/lateral translation

SECONDARY OUTCOMES:
Mean operation time | Time when the operation was begun

CONTACTS AND LOCATIONS:
Overall Officials: Yu Zhang, PhD, Study Chair — Hospital of Orthopedics, Guangzhou General Hospital of Guangzhou Military Command, 111 Liuhua Road, Guangzhou 510010, China

IPD SHARING:
Plan to Share IPD: No